CLINICAL TRIAL: NCT01645787
Title: Columbia SMA Project: 4-AP as a Potential SMA Therapeutic Agent and Biological Mechanisms of Action
Brief Title: Short and Long Term Treatment With 4-AP in Ambulatory SMA Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Claudia Chiriboga, Professor of Neurology and Pediatrics at CUMC, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAI7400
Record Dates: First submitted 2012-07-05; First posted 2012-07-20 (Estimated); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; 4-aminopyridine; dalfampridine; Ampyra
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — 4-Aminopyridine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4-aminopyridine (Ampyra) (Active Comparator): 10 mg tab/ 1 tab twice daily
  Interventions: Drug: 4-aminopyridine
- Sugar pill (Placebo Comparator): Placebo 1 tab /twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 4-aminopyridine — 10 mg/twice daily
  Other Names: dalfampridine-ER; Ampyra
  Arms: 4-aminopyridine (Ampyra)
Drug: Placebo — Crossover study involving one trial with sugar pill (placebo)
  Other Names: Sugar pill
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to assess whether 4-AP (Dalfampridine-ER, Ampyra) improves walking ability and endurance in adult patients with Spinal muscular atrophy (SMA) Type 3 compared to placebo and whether the duration of treatment affects outcome.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a genetically determined neuromuscular disorder that results in muscle weakness and impaired functional mobility. Fatigue is a common symptom in SMA with a resultant impact on physical function and quality of life however the precise mechanisms are unknown. At present there is no treatment for SMA. There is evidence that 4-AP improves function in SMA animal models. In patients with multiple sclerosis, 4-AP was found to improve walking ability and diminish fatigue. The purpose of the study is to determine whether treatment with 4-AP is associated with an increase in walking speed and endurance compared to placebo and whether the duration of treatment affects outcome. The study comprises a short term treatment trial in which participants are treated for 2 weeks with 4-AP and placebo in random sequence followed by a long treatment trial of 6 weeks in which patients are also treated with placebo and 4 AP. The primary outcome measure of the clinical study will be the six minute walk test (6MWT), which has been documented to be a valid and sensitive instrument to identify fatigue among ambulatory SMA patients. We will also assess the effect of 4-AP on muscle and nerve electrical function via electromyography (EMG) during the short term trial. Results of this study may provide support for larger clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 50 years at the time of enrollment
2. Have genetically confirmed SMA 3 (homozygous absence of SMN1 exon 7)
3. Ability to walk at least 25 meters without assistance
4. Be free of major orthopedic deformities (i.e. scoliosis, contractures)
5. Normal Cystatin C clearance (> 80 ml/min)

Exclusion Criteria:

1. Patients with a history of seizures
2. Patients with any renal impairment
3. Inability to comply with the study procedures
4. Unstable medical illness
5. Any ventilatory assistance
6. Taking experimental medication for SMA other than under this protocol
7. Pregnancy or lactation
8. Menstruating women, not sterilized or not using effective birth control
9. Planning to undergo scoliosis surgery within the next 10 months
10. Inability to give informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia A. Chiriboga, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- 4-aminopyridine, Then Placebo: Participants first received 4-aminopyridine 10 mg/twice daily for two weeks. After a washout period of one week, they then received placebo tablet (matching 4-aminopyridine) twice daily for two weeks (short term study).
  After a washout period of two weeks (following short term study), participants received 4-aminopyridine 10 mg/twice daily for six weeks. After a washout period of two weeks, they then received placebo tablet (matching 4-aminopyridine) twice daily for six weeks (long term study).
- Placebo, Then 4-aminopyridine: Participants first received placebo tablet (matching 4-aminopyridine) twice daily for two weeks. After a washout period of one week, they then received 4-aminopyridine 10 mg/twice daily for two weeks (short term study).
  After a washout period of two weeks (following short term study), participants first received placebo tablet (matching 4-aminopyridine) twice daily for six weeks. After a washout period of two weeks, they then received 4-aminopyridine 10 mg/twice daily for six weeks (long term study).
Period: First Intervention Short Term (2 Weeks)
Arm/Group | 4-aminopyridine, Then Placebo | Placebo, Then 4-aminopyridine
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | 4-aminopyridine, Then Placebo | Placebo, Then 4-aminopyridine
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | 4-aminopyridine, Then Placebo | Placebo, Then 4-aminopyridine
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | 4-aminopyridine, Then Placebo | Placebo, Then 4-aminopyridine
Started | 6 | 5
Completed | 5 | 5
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Third Intervention Long Term (6 Weeks)
Arm/Group | 4-aminopyridine, Then Placebo | Placebo, Then 4-aminopyridine
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | 4-aminopyridine, Then Placebo | Placebo, Then 4-aminopyridine
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Fourth Intervention (6 Weeks)
Arm/Group | 4-aminopyridine, Then Placebo | Placebo, Then 4-aminopyridine
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 11 subjects have thus been consented/enrolled in the study: 11 completed the short term component and 10 completed the long term components, a figure corresponding to the original targeted complement of the long term component.
Groups:
- All Subjects: Includes all subjects who had been consented/enrolled and completed the short term component of the study.
Arm/Group | All Subjects
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 37.7 [20 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Six Minute Walk Test (6MWT) With Kinematic Evaluation of Gait (Short Term)
Description: The primary outcome measure will be distance walked in the 6MWT. This measure is an objective evaluation of functional capacity which measures the distance a person can walk quickly in six minutes and is most representative of a person's ability because the test intensity is self-selected. The 6MWT can be safely performed in ambulatory SMA patients and correlates with standard SMA outcome measures including timed walking tests. In SMA, the 6MWT may be more sensitive to clinically meaningful changes in patients with type 3 SMA as it is a direct measure of their functional mobility.
Time Frame: Day 14 of each short-term intervention period
Measure: Mean (90% Confidence Interval); unit: meters
Groups:
- Short Term 4-aminopyridine (Ampyra): Participants who received 4-aminopyridine 10 mg/twice daily for two weeks.
- Short Term Placebo: Participants who received placebo twice daily (matching 4-aminopyridine) for two weeks.
Arm/Group | Short Term 4-aminopyridine (Ampyra) | Short Term Placebo
Number analyzed (Participants) | 11 | 11
meters | 293.05 [233.60 to 352.50] | 299.50 [240.05 to 358.95]

2. Primary Outcome: Six Minute Walk Test (6MWT) With Kinematic Evaluation of Gait (Long Term)
Description: as for outcome 1
Time Frame: Day 42 of each long-term intervention period
Population: Ten of 11 participants completed the long term study. One participant withdrew prior to the long term study due to worsening migraine.
Measure: Mean (90% Confidence Interval); unit: meters
Groups:
- Long Term 4-aminopyridine (Ampyra): Participants who received 4-aminopyridine 10 mg/twice daily for six weeks.
- Long Term Placebo: Participants who received placebo twice daily (matching 4-aminopyridine) for six weeks.
Arm/Group | Long Term 4-aminopyridine (Ampyra) | Long Term Placebo
Number analyzed (Participants) | 10 | 10
meters | 299.10 [235.93 to 362.27] | 295.20 [232.03 to 358.37]

3. Secondary Outcome: Hammersmith Functional Motor Scale, Expanded (HFMSE) (Short Term)
Description: Assessments of motor function are clinically relevant and are a good adjunct to tests of walking ability. The HFMSE, a 33-item scale designed for SMA type 2 and 3 patients, and is associated with minimal patient burden requiring only standard equipment and is completed on average in less than 15 minutes. The HFMSE showed good test-retest reliability and is correlated with other clinical and physiological measures in SMA. The score range is 0 (all items failed) to 66 (all items achieved unaided), with higher score indicating higher level of motor function.
Time Frame: Day 14 of each short-term intervention period
Measure: Mean (90% Confidence Interval); unit: score
Groups:
- Short Term 4-aminopyridine (Ampyra): Participants who received 4-aminopyridine (Ampyra) 10mg/twice daily for two weeks.
- Short Term Placebo: Participants who received placebo (matching 4-aminopyridine) twice daily for two weeks.
Arm/Group | Short Term 4-aminopyridine (Ampyra) | Short Term Placebo
Number analyzed (Participants) | 11 | 11
score | 50.84 [48.53 to 53.16] | 50.43 [48.11 to 52.74]

4. Secondary Outcome: Hammersmith Functional Motor Scale, Expanded (HFMSE) (Long Term)
Description: as for outcome 3
Time Frame: Day 42 of each long-term intervention period
Population: as for outcome 2
Measure: Mean (90% Confidence Interval); unit: score
Arm/Group | Long Term 4-aminopyridine (Ampyra) | Long Term Placebo
Number analyzed (Participants) | 10 | 10
score | 50.90 [48.49 to 53.31] | 50.30 [47.89 to 52.71]

5. Secondary Outcome: Manual Muscle Testing (MMT) Total Score (Short Term)
Description: MMT will involve pushing and pulling against the evaluators hand (MMT). The purpose of this test is to measure the strength in different muscles. MMT was performed on 28 muscle groups (8 muscle groups on each leg and 6 muscle groups on each arm), including proximal and distal musculature. The score range for each muscle group is 0 to 10, with a higher score indicating better muscle strength. The total score range is 0 to 280.
Time Frame: Day 14 of each short-term intervention period
Measure: Mean (90% Confidence Interval); unit: score
Arm/Group | Short Term 4-aminopyridine (Ampyra) | Short Term Placebo
Number analyzed (Participants) | 11 | 11
score | 181.86 [170.50 to 193.23] | 182.23 [170.86 to 193.59]

6. Secondary Outcome: Manual Muscle Testing (MMT) Total Score (Long Term)
Description: as for outcome 5
Time Frame: Day 42 of each long-term intervention period
Population: as for outcome 2
Measure: Mean (90% Confidence Interval); unit: score
Arm/Group | Short Term 4-aminopyridine (Ampyra) | Short Term Placebo
Number analyzed (Participants) | 10 | 10
score | 177.80 [163.85 to 191.75] | 181.10 [167.15 to 195.05]

7. Secondary Outcome: Motor Unit Number Estimation (MUNE)
Description: Motor Unit Number Estimation (MUNE) is a noninvasive test that identifies the number of motor units (motor nerve cells and the territory of muscle fibers they control) using electrical muscle stimulation and recording the response. The nerve conduction study involves the administration of modest electrical stimulations (pulsations or throbbing sensations from low level electricity) to a total of 4 nerves in the right arm and leg while recording the response over a muscle innervated by each nerve. MUNE is calculated by determining the compound motor action potential (CMAP) amplitude or area under the curve of a distal muscle in response to supramaximal stimulation, and then dividing the result by the amplitude or area under the curve of a single motor unit action potential.
Time Frame: Day 14 of each short-term intervention period
Population: MUNE testing was conducted only during the short term study.
Measure: Mean (90% Confidence Interval); unit: motor units
Arm/Group | Short Term 4-aminopyridine (Ampyra) | Short Term Placebo
Number analyzed (Participants) | 11 | 11
motor units | 190.86 [142.16 to 239.56] | 194.26 [145.30 to 243.23]

ADVERSE EVENTS:
Time Frame: 5 weeks for Short Term study, 16 weeks for Long Term study (up to 21 weeks per participant)
Groups:
- 4-aminopyridine (Short Term); 4-aminopyridine (Long Term): Participants who received 4-aminopyridine 10 mg/twice daily
- Placebo (Short Term); Placebo (Long Term): Participants who received placebo (matching 4-aminopyridine) twice daily
Arm/Group | 4-aminopyridine (Short Term) | Placebo (Short Term) | 4-aminopyridine (Long Term) | Placebo (Long Term)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 9/11 | 4/11 | 11/11 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 4-aminopyridine (Short Term) (N=11) | Placebo (Short Term) (N=11) | 4-aminopyridine (Long Term) (N=11) | Placebo (Long Term) (N=10)
Upset Stomach (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (General disorders) | 0 | 1 | 0 | 1
Fall (General disorders) | 2 | 2 | 6 | 1
Dizziness (General disorders) | 3 | 0 | 2 | 0
Headache/migraine (General disorders) | 1 | 1 | 1 | 0
Tremors (General disorders) | 0 | 0 | 1 | 0
Upper Respiratory Infection (URI) (Infections and infestations) | 1 | 0 | 1 | 1
Insomnia (General disorders) | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes